CLINICAL TRIAL: NCT06362330
Title: Knowledge-guided Causal Diagnostic Network for the Detection of Muscle-invasive Bladder Cancer With Single T2-weighted Imaging
Brief Title: Multi-parametric MRI in Patients of Bladder Cancer
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-SR-471
Record Dates: First submitted 2024-04-06; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Muscle-invasive Bladder Cancer; Artificial Intelligence
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- muscle-invasive bladder cancer: The postoperative pathology was muscle-invasive bladder cancer
  Interventions: Other: magnetic resonance imaging
- non-muscle-invasive bladder cancer: The postoperative pathology was non-muscle-invasive bladder cancer
  Interventions: Other: magnetic resonance imaging

INTERVENTIONS:
Other: magnetic resonance imaging — Patients of bladder cancer underwent multiparameter magnetic resonance imaging before surgery

SUMMARY:
Accurate preoperative detection of muscle-invasive bladder cancer remains a clinical challenge. The investigators aimed to develop and validate a knowledge-guided causal diagnostic network for the detection of muscle-invasive bladder cancer with multiparametric magnetic resonance imaging(MRI).

DETAILED DESCRIPTION:
Patients who underwent bladder MRI were retrospectively collected at three centers between January 2013 and September 2023. The investigators first constructed a nnUNet to segment causal region where muscle-invasive bladder cancer may occur. Subsequently, the investigators explored a causal network based on a modified ResNet3d-18 by striking a fine balance between nnUNet awareness and a self-supervised learning (SSL) model, which steered model to emulate diagnostic acumen of expert in staging muscle-invasive bladder cancer at MRI. Model was trained in center 1, and independently tested in center 1, center 2 and center 3. Ablation test was performed among all 13 Ablation-Test models using either single or multi-parametric MRI. Benefit was tested in six radiologists using vesical imaging-reporting and data system (VI-RADS) versus network-adjusted VI-RADS.

ELIGIBILITY:
Inclusion Criteria:

* Urothelial carcinoma of the bladder confirmed by final histopathology ②Received a standard contrast-enhanced 3.0T mpMRI before surgery ③All tumors within patients included were resected and received pathologic examination separately

Exclusion Criteria:

①Absence of surgical interventions

②With inadequate image quality or with inadequate pathology for analysis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Preoperative multi-parameter magnetic resonance imaging is essential to ascertain whether patients with bladder cancer exhibit muscular invasion, facilitating the selection of appropriate treatment options.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Muscle-invasive bladder cancer | one month
  The artificial intelligence diagnosis results, based on preoperative MRI, indicated muscle-invasive bladder cancer. Subsequently, this preoperative diagnosis was compared with the postoperative pathological diagnosis to evaluate the diagnostic performance of the artificial intelligence.
Non-muscle-invasive bladder cancer | one month
  The artificial intelligence diagnosis results, based on preoperative MRI, indicated non-muscle-invasive bladder cancer. Subsequently, this preoperative diagnosis was compared with the postoperative pathological diagnosis to evaluate the diagnostic performance of the artificial intelligence.

CONTACTS AND LOCATIONS:
Locations (1):
- Yu-Dong Zhang, Nanjing, China